CLINICAL TRIAL: NCT01837303
Title: chemQbiosciences:Manual Liquid Based Cytology
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 13-1341
Record Dates: First submitted 2013-04-08; First posted 2013-04-23 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-04

CONDITIONS: Cervical Dysplasia; Cervical Cancer
Keywords: Cervical dysplasia; Cervical cancer
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms | interventions — Papanicolaou Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liquid based cytology: All participants will undergo both manual and conventional automated liquid based cytology (pap smear, cervical cytology).
  Interventions: Procedure: Pap smear

INTERVENTIONS:
Procedure: Pap smear — A pap smear/cervical cytology is performed using a spatula and brush to obtain cells from the ectocervical and endocervical region of the cervix. The specimen will be collected twice to put in the standard clinical pap medium and another to put in the study pap medium.
  These slides will be processed so that they may be reviewed by a single board certified pathologist.
  There are no other interventions or follow up. All participants will undergo the above described procedures. There is no placebo.
  Other Names: cervical cytology

SUMMARY:
Purpose: To assess equivalence between low cost manual liquid based cytology (pap smear) and standard Thin prep cytology screening.

Participants: 100-120 healthy women presenting for standard pap smear screening

Procedures (methods): After routine care pap smear, another pap smear will be performed and placed in the study medium. Clinical care pap and study pap will be reviewed by a single pathologist to assess for equivalent findings.

Hypothesis: Manual liquid based cytology is equivalent to conventional liquid based cytology.

DETAILED DESCRIPTION:
Purpose: To assess equivalence between low cost manual liquid based cytology (pap smear) and standard Thin prep cytology screening.

Participants: 100-120 healthy women presenting for standard pap smear screening

Procedures (methods): After routine care pap smear, another pap smear will be performed and placed in the study medium. The study pap medium will be processed using the manufacturers instructions and then clinical care pap and study pap will be reviewed by a single pathologist to assess for equivalent findings.

ELIGIBILITY:
Inclusion Criteria:

* Female ages 18 years or older
* English speaking
* Presenting for pap smear examination

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 76 healthy women presenting for standard pap smear screening
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Compare cytologic outcomes using manual liquid based cytology to conventional | 4 months
  A single board certified Pathologist will blindly review the study pap smear and clinical pap smear. There results will be compared for differences.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Rahangdale, MD, MPH, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina Hospitals, Chapel Hill, North Carolina, United States